CLINICAL TRIAL: NCT01210404
Title: Open Label Single Sequence Study To Estimate The Effect Of Filibuvir (PF-00868554) On S-And R-Methadone In Subjects Receiving Chronic Methadone Treatment And To Evaluate The Pharmacokinetics Of Filibuvir
Brief Title: Drug Interaction Study Of Filibuvir With Methadone Among Subjects On Chronic Methadone Maintenance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8121023
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis C
Keywords: Drug interaction with methadone.
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — filibuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1.0 (Experimental)
  Interventions: Drug: filibuvir

INTERVENTIONS:
Drug: filibuvir — Filibuvir, 600mg bid administered along with methadone on days 2-11

SUMMARY:
Filibuvir, a CYP3A4 inhibitor is being developed for the treatment of chronic Hepatitis C infection. Given the likelihood of co administration of filibuvir and methadone, this study will evaluate the effect of filibuvir on the pharmacokinetics of R/S Methadone.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, without evidence of infection with HIV,HBV or HCV, who are on chronic methadone maintenance for at least three months and at a stable dose for at least 1 week prior to study start.

Exclusion Criteria:

* Evidence of chronic diseases including HIV, HBV or HCV.
* Evidence of acute or chronic liver disease.
* Treatment with prescription or nonprescription drugs other than methadone within 7 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Methadone plasma pharmacokinetic parameters, AUC24, Cmax | day 1
Methadone plasma pharmacokinetic parameters, AUC24, Cmax | day 11

SECONDARY OUTCOMES:
Methadone plasma pharmacokinetic parameters Tmax and C24h | day 1
Methadone plasma pharmacokinetic parameters Tmax and C24h | day 11
Filibuvir plasma pharmacokinetic parameters: Auc 12, Cmax, and Tmax. | day 2
Filibuvir plasma pharmacokinetic parameters: Auc 12, Cmax, and Tmax. | day 11
Safety and tolerability, including adverse events, vital signs, 12 lead ECG and lab safety assessments. | days 0-12
Symptoms of methadone withdrawal as assessed by short Opiate Withdrawal Scale, Desires for Drug questionnaire and pupillary diameter measurement . | days 0-12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8121023&StudyName=Drug%20Interaction%20Study%20Of%20Filibuvir%20With%20Methadone%20Among%20Subjects%20On%20Chronic%20Methadone%20Maintenance